CLINICAL TRIAL: NCT06455696
Title: Intra-Hospital Transport of Critically Ill Patients in Intensive Care Unit
Acronym: TIGRHOU
Status: Recruiting | Type: Observational
Sponsor: French Society for Intensive Care (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00866-39
Record Dates: First submitted 2024-05-27; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Critical Illness; Transportation Accidents; Intensive Care Unit
Keywords: Intra-hospital transport; Critical ill patients; Intensive care unit
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intra-hospital transport is a frequent procedure in the ICU, involving patients with the highest severity scores. Although some studies estimate the rate of adverse events to be around 33% during intra-hospital transport, including 4% of serious adverse events, the epidemiological data available is small, heterogeneous, and probably subject to methodological bias.

The aim of this study observational prospective observatoinal study is to determine:

* the different practices existing between ICUs ("practice survey")
* the occurrence of adverse events during intra-hospital transport provided by intensive care units (epidemiological study)

DETAILED DESCRIPTION:
This is a multicenter prospective observational study on evaluation of practices between ICUs and to describe the occurence of adverse events during intra-hospital transport provided by ICUs (epidemiological study)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old
* Hospitalized in ICU
* Requiring an intra-hospital transport (e.g imagery, operating room, etc) by the ICU team
* With a departure from ICU and arrival to ICU

Exclusion Criteria:

* Person under guardianship
* Protected Majors
* Already included in the study
* Transport for an ICU discharge in a medical or surgical ward
* Transport with another team than the ICU team
* Not affiliated to French social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized in an ICU and requiring an intra-hospital transport with a departure from ICU and arrival to ICU will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 645 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events during intra-hospital transport in critical ill patients managed by an ICU team | During the intra-intrahospital transport [maximum 3 hours]
  The number of adverse events during intra-hospital transport managed by an ICU team, as a proportion of the number of transports performed.

SECONDARY OUTCOMES:
Incidence of non-serious adverse events occurring during intra-hospital transport. | During the intra-intrahospital transport [maximum 3 hours]
  3) Rate of types of (non-serious) adverse events occurring during intra-hospital transport including O Rate of Withdrawal or mobilization of equipment with low risk of serious complication (e.g. VVP withdrawal, urinary catheter, nasogastric tube, mobilization of endotracheal tube without extubation) O Rate of Non-severe hemodynamic failures (occurrence of arterial hypotension with MAP between 40 and 65 mmHg, or catecholamine increase < 10% during transport) O Rate of Non-severe respiratory failure (desaturation with a SpO2 ≥ 80%) O Rate of Metabolic failure (e.g. hypoglycemia on return from transport) O Rate of Neurological complications (consciousness disorders occurring without sedation, agitation) O Rate of Material failures (O2 or ventilator failure, electrical syringe pump failure)
Incidence of serious adverse events occurring during intra-hospital transport. | During the intra-intrahospital transport [maximum 3 hours]
  4) Rate of serious adverse events occurring during intra-hospital transport including O Death O Cardiorespiratory arrest O Accidental extubation and/or need for re-intubation, or removal of high-risk equipment (e.g. central venous catheter, arterial catheter, endotracheal tube) O Severe hemodynamic failure (arterial hypotension with MAP < 40 mmHg, introduction or increase of catecholamines ≥ 10% during transport) O Severe respiratory failure (desaturation with SpO2 < 80% or massive inhalation)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided